CLINICAL TRIAL: NCT04934007
Title: A Randomized Control Trial of Bilateral Lateral OFC rTMS in Obsessive Compulsive Disorder
Brief Title: Bilateral Lateral OFC rTMS in Obsessive Compulsive Disorder
Acronym: ORBITOC3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Henri Laborit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-A02544-49
Record Dates: First submitted 2021-06-07; First posted 2021-06-22 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: rTMS; D-B80 A/P
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active stimulation (Experimental): Active rTMS stimulation , 2 session per day during 10 days.
  Interventions: Device: rTMS Treatment
- Sham Stimulation (Sham Comparator): Sham rTMS stimulation , 2 session per day during 10 days.
  Interventions: Device: rTMS Treatment

INTERVENTIONS:
Device: rTMS Treatment — 1 Hz rTMS

SUMMARY:
According to the literature the lateral part of the Orbito Frontal Cortex (lOFC) is a relevant bilateral target for repetitive Trans-cranial Magnetic Stimulation (rTMS) in Obsessive Compulsive Disorder (OCD). Both hemispheres are concerned in terms of target.

ELIGIBILITY:
Inclusion Criteria:

* Age: Participants will be both males and females, 18-65 years of age included.
* diagnosis of OCD
* all the patients must have failed to respond to at least two different pharmacological treatment used for at least 6 weeks
* Affiliation to a social security system (recipient or assignee),
* Signed written inform consent form

Exclusion Criteria:

* The exclusion criteria are a diagnosis of another psychiatric disorder (except for anxious disorders), a diagnosis of a significant active medical illness, pregnancy or other neurological illness
* In accordance with the safety criteria for rTMS, patients with a history of seizure or bearing pacemakers, mobile metal implants, implanted medical pumps, or metal clips placed inside the skull will also be excluded
* The patients won't be allowed to change their medication during the trial. The treatment must be stable at least 3 week before day 0.
* Female subject who is pregnant, or of child-bearing age, sexually active and not using reliable contraception or who is nursing,
* Patient under curators
* Patient hospitalized under duress
* Patient unable to give his or hers informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2021-09-06 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Yale Brown Obsessive Compulsive Scale score | baseline and 25 days
  Significant clinical change (≥ 25%) from baseline to two weeks after the treatment sequence, assessed by a significant reduction in YBOCS scores at day 25

SECONDARY OUTCOMES:
Yale Brown Obsessive Compulsive Scale | baseline and 70 days
  Significant clinical change of the YBOCS score (≥25% decrease), from baseline to day 70
general assessement functioning (GAF) | baseline and 25 days
  Change of the general assessement functioning (GAF) at day 25
general assessement functioning (GAF) | baseline and 70 days
  Change of the general assessement functioning (GAF) at day 70
Clinical Global Impression (CGI) | baseline and 25 days
  Clinical Global Impressions (CGI) change at day 25
Clinical Global Impression (CGI) | baseline and 70 days
  Clinical Global Impressions (CGI) change at day 70
Adverse events linked to the rTMS treatment | 70 days
  Number and types of adverse events linked to the rTMS treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ghina Harika-Germaneau, Study Director — Centre Hospitalier Henri Laborit
Locations (2):
- France (2):
  - Sorbonne University, Pitié-Salpêtrière Hospital, Paris
  - Centre Hospitalier Henri Laborit, Poitiers